CLINICAL TRIAL: NCT01865890
Title: Prevalence of Clopidogrel (Plavix) Resistance in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Suzanne El-Sayegh, Nephrology Attending, Assoc. Chair of Medicine, Northwell Health
Other Study IDs: 10-016
Record Dates: First submitted 2010-06-09; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Cardiovascular Disease
Keywords: Plavix or clopidogrel resistance
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient on hemodialysis taking plavix: patient on hemodialysis taking plavix

SUMMARY:
The investigators are trying to find out if Clopidogrel (Plavix) is as effective in hemodialysis patients as in patients not hemodialysed.

DETAILED DESCRIPTION:
Cardiovascular disease is very frequent in hemodialysis patients. Lot of hemodialysis patients are on Clopidogrel (plavix). Their is some evidence that clopidogrel is not effective in hemodialysis as it is effective in patient without kidney problem.

VerifyNow plavix is a machine that measure the ability of the blood to clot after giving plavix.

We will collect blood from hemodialysis patients on plavix and check the ability of their blood to clot and thus indirectly measuring the efficacy of Plavix.

ELIGIBILITY:
Inclusion Criteria:

* All patients on hemodialysis taking Plavix

Exclusion Criteria:

* known to have bleeding disorder
* Severely anemic with hemoglobin level (Hb) < 10g/dl
* Low Platelets < 10000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients who are taking plavix daily
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Prevalence Of Plavix resistance | 1 day ( one study visit)
  Plavix resistance is reported using the PRU values given by the VerifyNow machine. PRU is P2Y12 Reaction Units which is correlated with platelet aggregation.

SECONDARY OUTCOMES:
assess the risk factors for plavix resistance in the hemodialysis population | 1 day (one study visit)
  Coronary Artery Disease (CAD) is very common in dialysis patients. Treatment of CAD include medical therapy, stent placement and surgery. Since Plavix is a medication that is commonly used after stent placement, we would like to assess the efficacy of this medication in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne El-Sayegh, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States